CLINICAL TRIAL: NCT06152120
Title: Preparing Surrogates of Dementia Patients for In-the-moment Decision Making Through a Structured Advance Care Planning Intervention: A Mixed-methods Pilot Study
Brief Title: Preparing Surrogates of Dementia Patients Through an Advance Care Planning Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, YUEN Jacqueline Kwan Yuk, Clinical Assistant Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 20212481
Record Dates: First submitted 2023-11-21; First posted 2023-11-30 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-03

CONDITIONS: Dementia
Keywords: dementia; advance care planning
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Intervention Model Description: The investigators will use a sequential mixed-methods approach including a pilot randomized controlled trial using a quantitative study to evaluate the effects of a structured nurse-facilitated ACP intervention and a qualitative study to explore the perceptions of the family surrogates and the ACP nurse facilitator on the ACP intervention.
  Each patient-family dyad will be randomized in a 1:1 ratio to ACP intervention vs. usual care before the baseline interview.
Who Masked: Outcomes Assessor
Masking Description: Research staff will be blinded to the study arm when collecting data from family surrogates by telephone at follow up time-points. The study biostatistician will also be blinded to the allocation of the study arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ACP Intervention arm (Experimental): The intervention consists of two components:
  1. Palliative care needs assessment During the patient's hospitalization, the ACP nurse facilitator will conduct a palliative care needs assessment including assessment of patient's dementia severity (using the FAST scale), symptoms, clinical condition, nutritional and functional status, as well as psychosocial information.
  2. Structured nurse-facilitated post-discharge ACP consultations with use of video decisions aids
     * ACP consultation 1 (1-2 weeks post discharge)
     * Video decision aids (Between consultations 1 and 2)
     * ACP consultation 2 (2-3 weeks post discharge)
     * ACP consultation 3 (3-4 weeks post discharge), if needed
  At the completion of the ACP intervention, the ACP nurse facilitator may refer patients to the CGAT EOL program via the link nurse if fulfill the program criteria and agreed by the family surrogate(s).
  Interventions: Other: Nurse-facilitated advance care planning intervention
- Usual care arm (No Intervention): Patient and family surrogate dyads will receive usual hospital and post-discharge care. A publicly available information leaflet on advance care planning from the Hospital Authority's website will be given to control family surrogates after randomization. If a surrogate seeks assistance in discussing advance care planning, the research staff will advise the surrogate to speak with the patient's medical providers.

INTERVENTIONS:
Other: Nurse-facilitated advance care planning intervention — The intervention consists of two components:
  Component 1. Palliative care needs assessment - The research nurse will conduct a palliative care needs assessment and also review related information from the medical chart, which will enable the nurse to provide tailored information on the patient's illness, prognosis, and palliative care needs during subsequent ACP consultations.
  Component 2: Structured nurse-facilitated ACP consultations - The research nurse will conduct post-discharge ACP consultations with the family surrogate, with content that includes: assess readiness for discussions, introduce video decision aides to provide related ACP information and share examples of family surrogates with similar experiences.
  Arms: ACP Intervention arm

SUMMARY:
The goal of this clinical trial is to evaluate the effects of a nurse-facilitated post-discharge advance care planning intervention with family surrogates of dementia patients on outcomes that reflect the preparedness of surrogates in decision-making.

The main question it aims to answer is, whether the ACP intervention as compared with usual care will increase family surrogates' self-efficacy in surrogate decision-making and reduce their levels of distress, and increase patient comfort and reduce acute healthcare utilization at 2 and 6 months.

Participants will be randomized to ACP intervention vs. usual care.

1. patients of the Intervention group will be assessed on palliative care needs, and surrogates of the Intervention group will participate in 2-3 nurse-led ACP consultations;
2. surrogates of both intervention and control groups will complete 3 surveys at different time points during their participation of the study.

Researchers will compare the intervention group and control group to see any differences in:

1. surrogate preparedness for decision-making,
2. distress of surrogate and satisfaction with the care of loved one with dementia at the end-of-life,
3. enrolment in Community Geriatric Assessment Team end-of-life care program,
4. advanced care program documentation in medical record,
5. patient comfort at end-of-life,
6. hospitalizations in the last 6 months of life.

DETAILED DESCRIPTION:
In order to test the ACP interventions that aim to engage surrogates' participation in ACP and improve their preparedness for decision-making rather than on documentation of advance care plans alone, the research team has developed a pilot structured, nurse-facilitated post-discharge ACP intervention with the aim to improve surrogates' preparedness for in-the-moment decision-making.

It does so by incorporating best practices for ACP communication, drawing from prior work of the research team and existing literature, combined with a focus on developing surrogates' self-efficacy for decision-making guided by Bandura's Social Cognitive Theory.

This application aims to test the intervention's effects on surrogate outcomes (decision-making self-efficacy and distress), patient outcomes (patient comfort and healthcare utilization), as well as process outcomes (ACP documentation, end-of-life care discussions between family members, and enrolment in end-of-life care programs).

The research hypotheses to be tested are as follows: the investigators will test whether the ACP intervention as compared with usual care will increase family surrogates' self-efficacy in surrogate decision-making and reduce their levels of distress, and increase patient comfort and reduce acute healthcare utilization at 2 and 6 months.

ELIGIBILITY:
Dyads of patients with dementia admitted for an unplanned hospital admission and their family surrogate will be eligible for the study.

Inclusion Criteria of patients:

- Patient (a) at or above the age of 60 years old, (b) with diagnosis of dementia based on DSM-5 Criteria for Major Neurocognitive Disorder and Stage 6d or above on the Functional Assessment Staging Tool (FAST), (c) residing in a residential care home that is participating in Hospital Authority Enhanced Community Geriatric Assessment Team End-of-Life (CGAT EOL) Care program and (d) has an eligible family decision-maker.

Exclusion Criteria of patients:

- Patient with (i) prior completed advance directive, (ii) On tube feeding at the time of index admission, (iii) currently enrolled in an end-of-life care program or palliative care service, or (iv) with family members who lack consensus on the primary family surrogate decision-maker.

Inclusion Criteria of surrogates:

- Surrogate (a) at or above the age of 18 years old, (b) identified as the patient's next of kin or legal guardian who is the 'key decision maker' in hospital records, and (c) able to provide informed consent for him/herself and the patient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2023-06-15 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Modified Family Member Decision-Making Self-efficacy Scale (FDMSE) - Chinese version | Baseline, 2-month, 6-month
  This is a modified 17-item version of the FDMSE, a valid and reliable scale that quantifies a family member's confidence (0-100, where 100 = greatest self-efficacy) in end-of-life care decision-making for a loved one.
Family Distress in Advanced Dementia Scale (FDAD) Dementia Preparedness Subscale - Chinese version | Baseline, 2-month, 6-month
  The FDAD is a validated 21-item scale rated on a 1-5 scale, with higher scores indicating greater family distress. The scale assesses three domains of distress of family members of nursing home residents with dementia: Emotional Distress, Dementia Preparedness, and Clinician Relations. The Chinese version of the FDAD has high content validity (CVI = 0.95). It has good internal consistency (Cronbach's alpha 0.83) and moderate test-retest reliability (ICC = 0.64).
  We will use the 5-item Dementia Preparedness subscale to evaluate family distress associated with lack of knowledge of the course of dementia and surrogate medical decision making.

SECONDARY OUTCOMES:
End-of-life care discussions with other family members | Baseline, 2-month, 6-month
  The number of conversations which the surrogate has with other family members regarding end-of-life care decisions for the patient with advanced dementia.
Documentation of ACP discussions with medical providers | Baseline, 2-month, 6-month
  Information on the date of ACP discussion, type of clinician(s) involved, and care decisions in the Hospital Authority Clinical Management System.
Enrolment in Community Geriatric Assessment Team End-of-Life (CGAT EOL) care program | 2-month, 6-month
  Occurrence and date of new enrolment in the CGAT EOL care program in the Hospital Authority Clinical Management System.
Comfort Assessment in Dying with Dementia (CAD-EOLD) | 2-month, 6-month
  Measure of common symptoms and conditions to assess comfort of advanced dementia patients across 4 domains: Physical Distress, Emotional Distress, Well Being, and Dying Symptoms.
Unplanned hospital admissions and hospitalization days | 2-month, 6-month
  The number of unplanned hospital admissions and hospitalization days in public and private hospitals.

CONTACTS AND LOCATIONS:
Overall Officials: Jacqueline Yuen, Dr, Principal Investigator — The University of Hong Kong
Locations (1):
- The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No